CLINICAL TRIAL: NCT06000982
Title: A Comparison Study of Reduced Dose of Post-transplantation Cyclophosphamide (PTCy 40mg/kg) Versus Standard (PTCY 50mg/kg): a Multi-center Study for Halo-identical Donor Transplantation
Brief Title: Comparison of Different Dose of Post-transplantation Cyclophosphamide as Graft Versus Host Disease Prophylaxis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Clinical Research Center (Unknown)
Responsible Party: Principal Investigator, Jiong HU, Deputy director, department of hematology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PTCY40-50
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: GVHD
Keywords: graft versus host disease (GVHD); post-transplantation cyclophosphamide (PTCy); allogeneic stem cell transplantation; haplo-identical donor
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTCy-40 (Experimental): Patients receive 40mg/kg PTCY (day+3 and +4) with tacrolimus from day+5 and low-dose ATG of 2,5mg/kg 72 hours after documentation neutrophil engraftment.
  Interventions: Drug: PTCY
- PTCy-50 (Active Comparator): Patients receive 50mg/kg PTCY (day+3 and +4) with tacrolimus from day+5 and low-dose ATG of 2,5mg/kg 72 hours after documentation neutrophil engraftment.
  Interventions: Drug: PTCY

INTERVENTIONS:
Drug: PTCY — PTCY as 40mg/kg or 50mg/kg at day +3 and +4 for GVHD prophylaxis

SUMMARY:
Post-transplantation cyclophosphamide (PTCY) is considered as major graft versus host disease (GVHD) prophylaxis. In our previous study, the investigators demonstrated that the standard dose PTCY of 50mg/kg with tacrolimus and post-engrafted low-dose anti-thymoglobulin (ATG) achieved low incidence of acute GVHD. More recently, it has been shown that reduced dose of PTCY of 40mg/kg is considered with similar efficacy as GVHD prophylaxis, In this study, a multi-center randomized comparison is planned to evaluate the clinical outcome of GVHD prophylaxis of PTCy 40 versus 50.

DETAILED DESCRIPTION:
Post-transplantation cyclophosphamide (PTCY) is considered as major graft versus host disease (GVHD) prophylaxis. In our previous study, the investigators demonstrated that the standard dose PTCY of 50mg/kg with tacrolimus and post-engrafted low-dose anti-thymoglobulin (ATG) achieved low incidence of acute GVHD. In the clinical setting, reduced dose of PTCY (40mg/kg) was used for patients over 60 or with high HCT-CI and the overall incidence of acute GVHD was similar to PTCY 50mg/kg but chronic GVHD was slightly increased. To confirmed our observation, in this study, a prospective multiple-center randomized comparison is planned to evaluate the clinical outcomes of reduced dose of PTCY (40mg/kg) versus 50mg/kg as GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies
* Patients undergo allogeneic stem cell transplantation from haplo-identical donors
* Patents with informed consent provided

Exclusion Criteria:

* Patients with active infection ()bacteria, fungal or viral)
* Patients with liver, renal and cardiac dysfunction not suitable for undergoing allogeneic stem cell transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
acute GVHD (grade II-IV) | day 100
  clinical documentation of grade II-IV aGVHD

SECONDARY OUTCOMES:
Non-relapse mortality | 1 year
  Death without documentation of disease relapse or progression (bone marrow >5% or with extra medullary diseases)
chronic GVHD | 1 year
  incidence of patients with clinical documentation of chronic GVHD
overall survival | 1 year
  Event defined as death of any causes
Disease-free survival | 1 year
  Event defined as death of any causes and disease relapse or progression
Survival without relapse and moderate to severe GVHD | 1 year
  Rate of patients remain alive without disease relapse or progression (bone marrow blast >5% or extra medullary diseases) and without documentation of grade III-IV acute GVHD and moderate to severe chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: chun Wang, Study Director — Zhaxin Hospital, Go Broad Health Care
Locations (2):
- China (2):
  - Shenzhen People's Hospital, Shenzhen, GaungDong
  - Rui Jin Hospital, Shanghai, Shanghai Municipality